CLINICAL TRIAL: NCT01195077
Title: Could Dietary Algae Affect Immunity and Viral Counts in People With HIV?
Acronym: HIV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Dietary Algae and HIV
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: HIV Infections
Keywords: HIV; Dietary intervention; Algae; HIV progression; Algae specific kind
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Seaweed, Spirulina, Seaweed + Spirulina (Experimental): Randomized to:
  Arm 1: Seaweed. Ten capsules of .5 grams per capsule for a total of 10 grams per day.
  Arm 2: Spirulina: Ten capsules of .5 grams per capsule for a total of 10 grams per day.
  Arm 3: Seaweed: (2.5 grams) plus Spirulina (2.5 grams). Ten capsules of .5 grams per capsule for a total of 10 grams per day.
  Interventions: Other: seaweed, spirulina, seaweed + spirulina

INTERVENTIONS:
Other: seaweed, spirulina, seaweed + spirulina — Arm 1: Seaweed. Ten capsules of .5 grams per capsule for a total of 10 grams per day.
  Arm 2: Spirulina: Ten capsules of .5 grams per capsule for a total of 10 grams per day.
  Arm 3: Seaweed: (2.5 grams) plus Spirulina (2.5 grams). Ten capsules of .5 grams per capsule for a total of 10 grams per day.
  Spirulina: Ten capsules of .5 grams per capsule for a total of 10 grams per day.

SUMMARY:
Drawing inferences from epidemiologic studies of HIV/AIDS as well well as cell culture and animal studies of HIV inhibition by algae, we propose algal consumption as one unifying characteristic of countries with anomalously low rates. HIV/AIDS incidence and prevalence in Eastern Asia (<1/10,000 adults in Japan and Korea), compared to Africa (≈1/10 adults) strongly suggest that differences in IV drug use and sexual behavior are insufficient to explain the 1000-fold variation. Even in Africa, AIDS/HIV rates vary. Spirulina is part of the daily diet for many people living in Chad, where prevalence of HIV has remained at less than 4% for more than 20 years. Average daily algae consumption in Asia and Africa ranges between 1 to 2 tablespoons (3 - 13 grams).

HIV viral load is the main indicator of infection, however CD4 helper cell counts are most predictive of morbidity and mortality.We hypothesized that the consumption of algae could be important in diminishing the risk of HIV infection, and subsequent progression, possibly by enhancing the immune response.

DETAILED DESCRIPTION:
Twelve HIV+ patients not on antiretroviral therapy were clinically evaluated and enrolled in the three-week study. Subjects received 10 algae capsules/d. Laboratory tests of CD4 counts and HIV RNA were performed at baseline, week 1, week 2, and week 3, and then once a month. Six subjects continued for between 4 and 14 months. In addition to CD4 lymphocyte counts and viral loads, subjects were evaluated monthly for Complete Blood Counts (CBC), Liver profile, Basic Metabolic Panel, and some subjects were evaluated for thyroid function and cholesterol. All subjects completed standard HIV Quality of Life questionnaires at each clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HIV
* Able to swallow pills

Exclusion Criteria:

* Allergy to iodine/seafood
* Thyroid disease
* Not taking antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Dietary algae influence on CD4 helper cells and HIV viral load | Once a week for first 3 weeks, then once a month
  The first 6 subjects participated for 3 weeks. After analysis of the results, it was determined that there were no side effects and some indication of benefit. The next 6 subjects participated for up to 14 months.

SECONDARY OUTCOMES:
Would seaweed (Undaria) or spirulina or a combination of the two algae have more benefit? | Participants were randomized to one of 3 treatments.
  The combination of the 2 algae appeared to have more benefit. However, the sample size was too small to make conclusions.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Teas, Ph.D., Principal Investigator — University of South Carolina
Locations (1):
- Cancer Prevention and Control Program/University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- [Result] Trinchero J, Ponce NM, Cordoba OL, Flores ML, Pampuro S, Stortz CA, Salomon H, Turk G. Antiretroviral activity of fucoidans extracted from the brown seaweed Adenocystis utricularis. Phytother Res. 2009 May;23(5):707-12. doi: 10.1002/ptr.2723. PMID 19107862
- [Result] Damonte EB, Matulewicz MC, Cerezo AS. Sulfated seaweed polysaccharides as antiviral agents. Curr Med Chem. 2004 Sep;11(18):2399-419. doi: 10.2174/0929867043364504. PMID 15379705
- [Result] Pereira HS, Leao-Ferreira LR, Moussatche N, Teixeira VL, Cavalcanti DN, Costa LJ, Diaz R, Frugulhetti IC. Antiviral activity of diterpenes isolated from the Brazilian marine alga Dictyota menstrualis against human immunodeficiency virus type 1 (HIV-1). Antiviral Res. 2004 Oct;64(1):69-76. doi: 10.1016/j.antiviral.2004.06.006. PMID 15451181
- [Result] Cumashi A, Ushakova NA, Preobrazhenskaya ME, D'Incecco A, Piccoli A, Totani L, Tinari N, Morozevich GE, Berman AE, Bilan MI, Usov AI, Ustyuzhanina NE, Grachev AA, Sanderson CJ, Kelly M, Rabinovich GA, Iacobelli S, Nifantiev NE; Consorzio Interuniversitario Nazionale per la Bio-Oncologia, Italy. A comparative study of the anti-inflammatory, anticoagulant, antiangiogenic, and antiadhesive activities of nine different fucoidans from brown seaweeds. Glycobiology. 2007 May;17(5):541-52. doi: 10.1093/glycob/cwm014. Epub 2007 Feb 12. PMID 17296677
- [Result] Rechter S, Konig T, Auerochs S, Thulke S, Walter H, Dornenburg H, Walter C, Marschall M. Antiviral activity of Arthrospira-derived spirulan-like substances. Antiviral Res. 2006 Dec;72(3):197-206. doi: 10.1016/j.antiviral.2006.06.004. Epub 2006 Jun 30. PMID 16884788
- [Result] Buffa V, Stieh D, Mamhood N, Hu Q, Fletcher P, Shattock RJ. Cyanovirin-N potently inhibits human immunodeficiency virus type 1 infection in cellular and cervical explant models. J Gen Virol. 2009 Jan;90(Pt 1):234-43. doi: 10.1099/vir.0.004358-0. PMID 19088294
- [Result] Wang H, Ooi EV, Ang PO Jr. Antiviral activities of extracts from Hong Kong seaweeds. J Zhejiang Univ Sci B. 2008 Dec;9(12):969-76. doi: 10.1631/jzus.B0820154. PMID 19067465
- [Result] Artan M, Li Y, Karadeniz F, Lee SH, Kim MM, Kim SK. Anti-HIV-1 activity of phloroglucinol derivative, 6,6'-bieckol, from Ecklonia cava. Bioorg Med Chem. 2008 Sep 1;16(17):7921-6. doi: 10.1016/j.bmc.2008.07.078. Epub 2008 Jul 29. PMID 18693022
- [Result] Queiroz KC, Medeiros VP, Queiroz LS, Abreu LR, Rocha HA, Ferreira CV, Juca MB, Aoyama H, Leite EL. Inhibition of reverse transcriptase activity of HIV by polysaccharides of brown algae. Biomed Pharmacother. 2008 Jun;62(5):303-7. doi: 10.1016/j.biopha.2008.03.006. Epub 2008 Apr 4. PMID 18455359
- [Result] Gideon TP, Rengasamy R. Toxicological evaluation of fucoidan from Cladosiphon okamuranus. J Med Food. 2008 Dec;11(4):638-42. doi: 10.1089/jmf.2007.0127. PMID 19053854
- [Result] Paskaleva EE, Lin X, Duus K, McSharry JJ, Veille JC, Thornber C, Liu Y, Lee DY, Canki M. Sargassum fusiforme fraction is a potent and specific inhibitor of HIV-1 fusion and reverse transcriptase. Virol J. 2008 Jan 15;5:8. doi: 10.1186/1743-422X-5-8. PMID 18197976
- [Result] Paskaleva EE, Lin X, Li W, Cotter R, Klein MT, Roberge E, Yu EK, Clark B, Veille JC, Liu Y, Lee DY, Canki M. Inhibition of highly productive HIV-1 infection in T cells, primary human macrophages, microglia, and astrocytes by Sargassum fusiforme. AIDS Res Ther. 2006 May 25;3:15. doi: 10.1186/1742-6405-3-15. PMID 16725040
- [Result] Ahn MJ, Yoon KD, Kim CY, Kim JH, Shin CG, Kim J. Inhibitory activity on HIV-1 reverse transcriptase and integrase of a carmalol derivative from a brown Alga, Ishige okamurae. Phytother Res. 2006 Aug;20(8):711-3. doi: 10.1002/ptr.1939. PMID 16775811
- [Result] Ahn MJ, Yoon KD, Min SY, Lee JS, Kim JH, Kim TG, Kim SH, Kim NG, Huh H, Kim J. Inhibition of HIV-1 reverse transcriptase and protease by phlorotannins from the brown alga Ecklonia cava. Biol Pharm Bull. 2004 Apr;27(4):544-7. doi: 10.1248/bpb.27.544. PMID 15056863
- [Result] Simpore J, Zongo F, Kabore F, Dansou D, Bere A, Nikiema JB, Pignatelli S, Biondi DM, Ruberto G, Musumeci S. Nutrition rehabilitation of HIV-infected and HIV-negative undernourished children utilizing spirulina. Ann Nutr Metab. 2005 Nov-Dec;49(6):373-80. doi: 10.1159/000088889. Epub 2005 Oct 11. PMID 16219988
- [Result] Simpore J, Kabore F, Zongo F, Dansou D, Bere A, Pignatelli S, Biondi DM, Ruberto G, Musumeci S. Nutrition rehabilitation of undernourished children utilizing Spiruline and Misola. Nutr J. 2006 Jan 23;5:3. doi: 10.1186/1475-2891-5-3. PMID 16430775
- [Result] Yamani E, Kaba-Mebri J, Mouala C, Gresenguet G, Rey JL. [Use of spirulina supplement for nutritional management of HIV-infected patients: study in Bangui, Central African Republic]. Med Trop (Mars). 2009 Feb;69(1):66-70. French. PMID 19499738